CLINICAL TRIAL: NCT01402700
Title: Visi-Pro™ Balloon Expandable Iliac Study (VISIBILITY™ Iliac)
Brief Title: VISIBILITY™ Iliac Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-1000
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Peripheral Arterial Disease; Claudication
Keywords: Peripheral arterial disease; claudication; stent; VISI-Pro; Iliac artery
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

ARMS (1):
- Visi-Pro™ Balloon Expandable Stent System (Experimental): The objective of the study is to confirm the safety and effectiveness of the Visi-Pro stent in the treatment of stenotic, restenotic or occluded lesions in the common and external iliac artery.
  Interventions: Device: Visi-Pro™ Balloon Expandable Stent System

INTERVENTIONS:
Device: Visi-Pro™ Balloon Expandable Stent System — Implantation of one or more study devices in the common and/or external iliac artery.

SUMMARY:
The VISIBILITY Iliac study is a prospective, multi-center, non-randomized study confirming the safety and effectiveness of stenting using the Visi-Pro™ Balloon Expandable Stent System for the treatment of stenotic, restenotic or occluded lesions in the common and external iliac artery.

ELIGIBILITY:
Inclusion Criteria:

* Patient has claudication as defined by a Rutherford Clinical Category Score of 2, 3 or 4.
* Evidence of ≥ 50% stenosis, restenosis or occlusion of target lesion(s) located in the common iliac artery and/or external iliac artery.
* Willing to comply with all follow-up evaluations at the specified times.
* Provides written informed consent prior to enrollment in the study.

Exclusion Criteria:

* Previous implantation of stent(s) in the target vessel.
* Received endovascular treatment of the target lesion within six months prior to the index procedure.
* Known hypersensitivity to contrast material that cannot be adequately pretreated.
* Known hypersensitivity to 316L stainless Steel.
* Life expectancy of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter L. Faries, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai; John H. Rundback, M.D., Principal Investigator — Holy Name Medical Center
Locations (1):
- Holy Name Medical Center, Teaneck, New Jersey, United States

REFERENCES:
- [Derived] Rundback JH, Peeters P, George JC, Jaff MR, Faries PL. Results From the VISIBILITY Iliac Study: Primary and Cohort Outcomes at 9 Months. J Endovasc Ther. 2017 Jun;24(3):342-348. doi: 10.1177/1526602817692960. Epub 2017 Feb 1. PMID 28351204

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Visi-Pro™ Balloon Expandable Stent System
Started | 75
Completed | 68
Not Completed | 7
Not completed — Death | 3
Not completed — Withdrawal by Subject | 3
Not completed — Missed Visit | 1

BASELINE CHARACTERISTICS:
Arm/Group | Visi-Pro™ Balloon Expandable Stent System
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Event Rate at 9 Months
Description: The Major Adverse Event rate at 9 months is defined as a composite of periprocedural death, in-hospital MI, clinically-driven target lesion revascularization and amputation of the treated limb through 9 months postprocedure.
Time Frame: 9 months
Measure: Number; unit: percentage of participants
Arm/Group | Visi-Pro™ Balloon Expandable Stent System
Number analyzed (Participants) | 75
percentage of participants | 4.0

ADVERSE EVENTS:
Time Frame: All events that occured within 9 months
Arm/Group | Visi-Pro™ Balloon Expandable Stent System
Serious Adverse Events (participants affected / at risk) | 38/75
Other Adverse Events (participants affected / at risk) | 22/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Visi-Pro™ Balloon Expandable Stent System (N=75)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1)
Catheter site haematoma (General disorders) | 5 (5)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic occlusion (Vascular disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Pleuropericarditis (Cardiac disorders) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Puncture site haemorrhage (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 4 (6)
Cellulitis (Infections and infestations) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Wound infection (Immune system disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 1 (2)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (2)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arterial spasm (Vascular disorders) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 3 (3)
Hypertensive crisis (Vascular disorders) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 5 (5)
Peripheral embolism (Vascular disorders) | 1 (1)
Subclavian steal syndrome (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Visi-Pro™ Balloon Expandable Stent System (N=75)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Oedema peripheral (General disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and Sponsor [or its agents] that restricts PI's rights to discuss or publish trial results without permission of the Sponsor.

Trial is still ongoing.